CLINICAL TRIAL: NCT00003869
Title: Phase III Randomized, Double-Blind Study of CAI and Placebo in Patients With Advanced Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Carboxyamidotriazole in Treating Patients With Stage III or Stage IV Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCI-2012-02898; NCI-2012-02898 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000067033; 97-24-51 (Other: North Central Cancer Treatment Group); NCCTG-97-24-51 (Other: CTEP); U10CA025224 (NIH)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Results first posted 2010-12-22 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2012-12

CONDITIONS: Stage IIIA Non-small Cell Lung Cancer; Stage IIIB Non-small Cell Lung Cancer; Stage IV Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — carboxyamido-triazole

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Arm I (CAI) (Experimental): Patients receive oral carboxyamidotriazole daily.
  Interventions: Drug: carboxyamidotriazole; Procedure: quality-of-life assessment; Other: laboratory biomarker analysis
- Arm II (placebo) (Placebo Comparator): Patients receive oral placebo daily
  Interventions: Other: placebo; Procedure: quality-of-life assessment; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: carboxyamidotriazole — Given PO
  Other Names: CAI; carboxyamido-triazole; carboxyaminoimidazole
  Arms: Arm I (CAI)
Other: placebo — Given PO
  Other Names: PLCB
  Arms: Arm II (placebo)
Procedure: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Randomized phase III trial to determine the effectiveness of carboxyamidotriazole in treating patients who have stage III or stage IV non-small cell lung cancer. Chemotherapeutic agents are modestly effective for the treatment of advanced lung cancer, with rapid tumor relapse and growth even after initial response to therapy. It is not yet known whether carboxyamidotriazole is more effective than no further treatment after standard chemotherapy for non-small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether oral administration of the carboxyaminoimidazole (CAI) is more effective than placebo in prolonging the overall survival in patients with non-small cell lung cancer stage III or stage IV non-small cell lung cancer who have been stable or had tumor regression following chemotherapy.

SECONDARY OBJECTIVES:

I. To evaluate the safety and tolerability of oral CAI following chemotherapy. II. To determine whether CAI prolongs time-to-disease progression relative to a placebo.

III. To evaluate whether a substantive effect in quality of life (QOL) can be detected between the CAI and placebo groups using the FACT-L and the UNISCALE.

IV. To document the response rate to CAI in patients with measurable or evaluable disease.

TERTIARY OBJECTIVES:

I. To evaluate genotypes at GSH-related loci as predictors of overall survival.

OUTLINE: This is a randomized, double-blind, multicenter study. Patients are stratified according to timing of first-line therapy (prior to registration vs after registration), disease stage (IIIA vs IIIB vs IV), therapy components (chemotherapy and thoracic radiotherapy vs chemotherapy only), ECOG performance status (0 vs 1 vs 2) and participating center. Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive oral carboxyamidotriazole daily.

ARM II: Patients receive oral placebo daily.

Treatment continues in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline and then monthly during study.

Patients are followed every 3 months for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* TRACK I: Histologically or cytologically confirmed NSCLC stage III or IV; disease must be stable or responding after standard chemotherapy (with or without TRT) for a minimum of 3 or a maximum of 6 months
* TRACK I: Not required to have measurable or evaluable disease at study entry
* TRACK I: Must have had one and only one prior chemotherapy regimen for NSCLC (radiosensitizers are allowed)
* TRACK I: =< 6 weeks from last dose of chemotherapy or TRT
* TRACK I: ECOG PS 0, 1, or 2
* TRACK I: ANC >= 1500/mm^3
* TRACK I: PLT >= 100,000/mm^3
* TRACK I: HgB >= 10.0 g/dL
* TRACK I: Total bilirubin =< 1.5 x UNL
* TRACK I: Alkaline phosphatase =< 3 x UNL
* TRACK I: AST =< 3 x UNL
* TRACK I: Creatinine =< 1.5 x UNL
* TRACK I: Expected survival of at least three months
* TRACK II AT REGISTRATION: Histologically or cytologically confirmed NSCLC stage III or IV
* TRACK II AT REGISTRATION: No prior chemotherapy for NSCLC
* TRACK II AT REGISTRATION: Expected survival of at least six months
* TRACK II AT REGISTRATION: Willingness to provide blood sample
* TRACK II AT RANDOMIZATION: STAB, PR, CR, REGR following 3-6 months of chemotherapy with or without radiation therapy
* TRACK II AT RANDOMIZATION: Must have had one and only one prior chemotherapy regimen for NSCLC (radiosensitizers are allowed)
* TRACK II AT RANDOMIZATION: =< 6 weeks from last dose of chemotherapy or TRT
* TRACK II AT RANDOMIZATION: ECOG PS 0, 1, or 2
* TRACK II AT RANDOMIZATION: ANC >= 1500/mm^3
* TRACK II AT RANDOMIZATION: PLT >= 100,000/mm^3
* TRACK II AT RANDOMIZATION: HgB >= 10.0 g/dL
* TRACK II AT RANDOMIZATION: Total bilirubin =< 1.5 x UNL
* TRACK II AT RANDOMIZATION: Alkaline phosphatase =< 3 x UNL
* TRACK II AT RANDOMIZATION: AST =< 3 x UNL
* TRACK II AT RANDOMIZATION: Creatinine =< 1.5 x UNL
* TRACK II AT RANDOMIZATION: Expected survival of at least three months

Exclusion Criteria:

* TRACK I: Pregnant, nursing women, females or sexual partners of childbearing potential not using adequate contraception (condoms, diaphragm, birth control pills, injections, intrauterine device [IUD], or abstinence, etc.) while on study treatment and for two months after discontinuing study treatment as this regimen may be harmful to a developing fetus or nursing child
* TRACK I: Untreated brain metastases
* TRACK I: Concomitant participation in a phase III lung cancer treatment trial
* TRACK I: Planned concurrent chemotherapy, immunotherapy or radiotherapy
* TRACK II AT RANDOMIZATION: Pregnant, nursing women, females or sexual partners of childbearing potential not using adequate contraception (condoms, diaphragm, birth control pills, injections, intrauterine device [IUD], or abstinence, etc.) while on study treatment and for two months after discontinuing study treatment as this regimen may be harmful to a developing fetus or nursing child
* TRACK II AT RANDOMIZATION: Untreated brain metastases
* TRACK II AT RANDOMIZATION: Planned concurrent chemotherapy, immunotherapy, or radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 1999-04; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edith Perez, Principal Investigator — North Central Cancer Treatment Group
Locations (1):
- North Central Cancer Treatment Group, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between April 1999 and January 2004, 194 patients were accrued to this study. This trial was closed to accrual prior to meeting the protocol projected 360 randomized patients due to slow accrual.
Pre-assignment Details: 186 patients were randomized to either arm
Groups:
- Carboxyamidotriazole: 250 mg carboxyamidotriazole administered daily
- Placebo: 250 mg placebo administered daily
Period: Overall Study
Arm/Group | Carboxyamidotriazole | Placebo
Started | 94 | 92
Completed | 53 | 80
Not Completed | 41 | 12
Not completed — Adverse Event | 14 | 3
Not completed — Withdrawal by Subject | 21 | 3
Not completed — Death | 1 | 2
Not completed — Alternative treatmnt, medical problems | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Carboxyamidotriazole | Placebo | Total
Number analyzed (Participants) | 94 | 92 | 186
Age, Customized [Number; unit: participants]
  <= 65 years | 37 | 50 | 87
  > 65 years | 57 | 42 | 99
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 37 | 79
  Male | 52 | 55 | 107
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 91 | 89 | 180
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Histology [Number; unit: participants]
  Bronchoalveolar/large cell | 6 | 13 | 19
  NOS (not otherwise specified) NSCLC/not avaliable | 16 | 11 | 27
  Adenocarcinoma | 51 | 55 | 106
  Squamous | 21 | 13 | 34
Eastern Cooperative Oncology Group Performance Score [Number; unit: Participants] — Classifies patients according to their functional impairment. Scores range from 0 (fully active) to 5 (death).
  Participants
    0 - Fully Active | 37 | 38 | 75
    1 - Ambulatory, restricted strenuous activity | 47 | 48 | 95
    2 - Ambulatory, unable to perform work activities | 10 | 6 | 16
Prior Response to Chemotherapy [Number; unit: participants]
  Complete | 5 | 4 | 9
  Partial | 38 | 45 | 83
  Regression | 9 | 8 | 17
  Stable | 42 | 35 | 77
Smoking Status [Number; unit: participants]
  Never | 11 | 10 | 21
  Former (quit >= 6 months) | 54 | 57 | 111
  Current | 20 | 15 | 35
  Not Reported | 9 | 10 | 19
TNM Stage [Number; unit: participants] — American Joint Committee on Cancer, Cancer Staging Manual http://www.cancerstaging.org/products/pasteditions.html
  participants
    IIIA/IIIB | 22 | 19 | 41
    IV | 72 | 73 | 145

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization to death of any cause. Participants who did not die or were lost to follow-up were censored at the time of last evaluation/follow-up date. Patients were followed for a maximum of 5 years from randomization. The median OS with 95%CI was estimated using the Kaplan Meier method.
Time Frame: up to 5 years
Population: Overall survival was analyzed on all randomized participants on an intent to treat basis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Carboxyamidotriazole | Placebo
Number analyzed (Participants) | 94 | 92
Months | 11.4 [9.2 to 13.9] | 10.5 [8.9 to 12.6]
Statistical Analysis 1: Comparison: Carboxyamidotriazole vs Placebo; Test type: Superiority or Other; p = 0.54, Log Rank

2. Secondary Outcome: Participants With Severe Non-hematologic Adverse Events
Description: Severe non-hematologic adverse events were defined as adverse events grade 3 or higher, regardless of attribution to study drug. Adverse events were graded according to the National Cancer Institute Common Toxicity Criteria (NCI CTC version 2.0)
Time Frame: every cycle during treatment
Population: All treated participants; all participants who received study treatment.
Measure: Number; unit: Participants
Arm/Group | Carboxyamidotriazole | Placebo
Number analyzed (Participants) | 90 | 92
Participants | 38 | 30
Statistical Analysis 1: Comparison: Carboxyamidotriazole vs Placebo; Test type: Superiority or Other; p = 0.18, Fisher Exact

3. Secondary Outcome: Time to Disease Progression (TTP)
Description: TTP is defined as the time from randomization to first documented disease progression(PD). Patients who were lost to follow-up were censored at the time of last evaluation. For patients who died without clear documentation, PD was assumed at the midpoint of the time interval between last evaluation and death. Median TTP was estimated using the Kaplan Meier method.
  Measurable PD: ≥25% increase in the sum of the products of two greatest perpendicular diameters of all indicator lesions or appearance of new lesion(s). Evaluable PD: definite increase in tumor size or appearance of new lesion(s)
Time Frame: up to 5 years
Population: TTP was analyzed on all randomized patients on an intent to treat basis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Carboxyamidotriazole | Placebo
Number analyzed (Participants) | 94 | 92
Months | 2.8 [2.1 to 3.8] | 2.4 [2.1 to 3.8]
Statistical Analysis 1: Comparison: Carboxyamidotriazole vs Placebo; Test type: Superiority or Other; p = 0.50, Log Rank

4. Secondary Outcome: Clinically Significant (10-point) Decrease in UNISCALE Quality of Life (QOL)Assessment From Baseline to Week 8
Description: The UNISCALE was used to assess QOL. UNISCALE is a single item global measure of QOL. Participant were to complete the questionnaire at baseline and every 8 weeks, prior to assessment by the treating physician. A high score indicates a higher quality of life while a low score represents a lower quality of life. A 10 point or greater decline (from baseline to week 8) in UNISCALE QOL score was considered clinically significant.
Time Frame: Baseline to week 8
Population: Participants who completed the baseline and week 8 UNISCALE assessment are included in the analysis.
Measure: Number; unit: participants
Arm/Group | Carboxyamidotriazole | Placebo
Number analyzed (Participants) | 39 | 63
participants | 28 [1.0 to 98.0] | 32 [0.7 to 100.0]
Statistical Analysis 1: Comparison: Carboxyamidotriazole vs Placebo; Test type: Superiority or Other; p = 0.04, Fisher Exact

5. Secondary Outcome: Clinically Significant (10-point) Decrease in Functional Assessment of Cancer Therapy for Lung Cancer (FACT-L) Quality of Life (QOL)Assessment From Baseline to Week 8
Description: The FACT-L is a 36-item Likert instrument that combines frequency of symptomatic/QOL problems with perceived relative importance of each issue. It includes 4 constructs of well being: physical, social/family, emotional and functional, and a fifth construct, additional concerns, dealing solely with tumor related symptoms. Questionnaires were completed at baseline and 8 weeks. Questions within each construct were summated to obtain a construct score. A higher score relates to higher quality of life. A 10 point or greater decline (from baseline to week 8) was considered clinically significant.
Time Frame: Baseline to week 8
Population: Participants who completed the baseline and week 8 FACT-L assessment are included in the analysis.
Measure: Number; unit: participants
Arm/Group | Carboxyamidotriazole | Placebo
Number analyzed (Participants) | 43 | 67
participants | 27 [40.2 to 93.1] | 33 [46.4 to 93.5]
Statistical Analysis 1: Comparison: Carboxyamidotriazole vs Placebo; Test type: Superiority or Other; p = 0.18, Fisher Exact

6. Secondary Outcome: Number of Patients With a Confirmed Tumor Responses Treated With CAI.
Description: Confirmed response was defined as a complete response (CR) or partial response (PR) for patients with measurable disease or as a CR or regression (REGR) for patients with evaluable disease noted on 2 consecutive evaluations at least 4 weeks apart.
  * CR: total disappearance of all tumor;
  * PR: >=50% reduction of the sum of the products of the two greatest perpendicular diameters of all indicator lesions;
  * REGR: Definite decrease in tumor size and no new lesion(s).
Time Frame: During Treatment (up to 5 years)
Population: This data was not (and will never be) analyzed as it was not submitted consistently due to the trial design. (Patients were required to be SD or better to be randomized to carboxyamidotriazole or placebo.)
Arm/Group | Carboxyamidotriazole | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Carboxyamidotriazole | Placebo
Serious Adverse Events (participants affected / at risk) | 9/90 | 6/92
Other Adverse Events (participants affected / at risk) | 87/90 | 84/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carboxyamidotriazole (N=90) | Placebo (N=92)
Arrythmia (Cardiac disorders) | 1 (1) | 0 (0)
Edema (Cardiac disorders) | 1 (1) | 0 (0)
Ischemia/Infarction (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular arrhythmias (SVT/atrial fibrillation/flutter) (Cardiac disorders) | 1 (1) | 0 (0)
Melena (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pain-Abdominal (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Fever-No ANC (General disorders) | 1 (1) | 0 (0)
Allergy (Immune system disorders) | 1 (1) | 0 (0)
Infection without neutropenia (Infections and infestations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Neuro-Sensory (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Adult respiratory distress syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Effusion-Pleural (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carboxyamidotriazole (N=90) | Placebo (N=92)
Anemia (Blood and lymphatic system disorders) | 44 (95) | 51 (151)
Blood/Bone Marrow (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Arrhythmia-Nodal (Cardiac disorders) | 1 (1) | 0 (0)
Arrythmia (Cardiac disorders) | 0 (0) | 2 (2)
Cardiovascular (Cardiac disorders) | 1 (1) | 0 (0)
Edema (Cardiac disorders) | 4 (4) | 8 (29)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular arrhythmias (SVT/atrial fibrillation/flutter) (Cardiac disorders) | 2 (2) | 2 (2)
Auditory (Ear and labyrinth disorders) | 0 (0) | 3 (6)
Inner Ear (Ear and labyrinth disorders) | 2 (6) | 1 (1)
Vision (Eye disorders) | 1 (1) | 0 (0)
Vision-Blurred (Eye disorders) | 6 (7) | 1 (1)
Vision-Double (Eye disorders) | 1 (1) | 0 (0)
Vision-Photopsia (Eye disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 14 (17) | 8 (14)
Diarrhea-BMT (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea-No Colostom (Gastrointestinal disorders) | 4 (4) | 4 (5)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dysphagia-esophageal related to radiation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 2 (4)
Gastrointestinal (Gastrointestinal disorders) | 0 (0) | 2 (4)
Hematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mouth Dryness (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 55 (102) | 28 (60)
Pain-Abdominal (Gastrointestinal disorders) | 3 (3) | 4 (6)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 3 (6)
Vomiting (Gastrointestinal disorders) | 29 (35) | 13 (17)
Fatigue (General disorders) | 48 (90) | 27 (52)
Fever-No ANC (General disorders) | 1 (1) | 1 (1)
Injection site reaction (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 5 (7) | 8 (11)
Pain-Chest (General disorders) | 3 (3) | 1 (1)
Rigors (General disorders) | 1 (1) | 2 (2)
Infection without neutropenia (Infections and infestations) | 4 (5) | 7 (7)
Alkaline phosphatase (Investigations) | 0 (0) | 8 (10)
Bilirubin (Investigations) | 2 (2) | 1 (1)
Creatinine (Investigations) | 8 (16) | 5 (9)
Leukopenia (Investigations) | 2 (2) | 5 (7)
Leukopenia-Peds (Investigations) | 0 (0) | 1 (1)
Lymphopenia (Investigations) | 3 (4) | 2 (5)
Metabolic/Lab (Investigations) | 0 (0) | 1 (7)
Neutropenia (Investigations) | 8 (9) | 7 (14)
Prothrombin Time (Investigations) | 1 (1) | 0 (0)
SGOT (AST) (serum glutamic oxaloacetic transaminase) (Investigations) | 3 (3) | 4 (6)
SGPT (ALT) (serum glutamic pyruvic transaminase) (Investigations) | 2 (2) | 2 (2)
Thrombocytopenia (Investigations) | 11 (12) | 10 (23)
Weight gain (Investigations) | 0 (0) | 1 (1)
Weight loss (Investigations) | 3 (4) | 4 (4)
Anorexia (Metabolism and nutrition disorders) | 28 (44) | 12 (15)
Bicarbonate (Metabolism and nutrition disorders) | 0 (0) | 1 (3)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (6) | 8 (18)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 4 (5)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 2 (4)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (7) | 7 (13)
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 10 (13)
Pain-Bone (Musculoskeletal and connective tissue disorders) | 2 (2) | 6 (7)
Pain-Tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 29 (43) | 15 (56)
CNS hemorrhage/bleeding (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 8 (9) | 6 (15)
Headache (Nervous system disorders) | 4 (6) | 7 (8)
Learning Disorder (Nervous system disorders) | 1 (1) | 0 (0)
Low Consciousness (Nervous system disorders) | 2 (2) | 0 (0)
Memory Loss (Nervous system disorders) | 2 (2) | 0 (0)
Neuralgia (Nervous system disorders) | 2 (4) | 1 (2)
Neuro-Motor (Nervous system disorders) | 4 (5) | 6 (10)
Neuro-Sensory (Nervous system disorders) | 53 (125) | 41 (163)
Seizure (Nervous system disorders) | 0 (0) | 2 (2)
Smell (Nervous system disorders) | 1 (1) | 0 (0)
Taste (Nervous system disorders) | 3 (4) | 3 (7)
Tremor (Nervous system disorders) | 1 (1) | 1 (6)
Vertigo (Nervous system disorders) | 0 (0) | 1 (4)
Anxiety (Psychiatric disorders) | 2 (2) | 4 (19)
Confusion (Psychiatric disorders) | 2 (2) | 1 (2)
Depression (Psychiatric disorders) | 5 (5) | 4 (7)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (2)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (2)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal (Renal and urinary disorders) | 0 (0) | 1 (3)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 1 (1)
Gynecomastia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 13 (22)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 15 (22) | 21 (49)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pain-Pleuritic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Voice Change (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 12 (16) | 15 (23)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (10)
Rash (Skin and subcutaneous tissue disorders) | 3 (4) | 4 (4)
Sweating (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Hot flashes (Vascular disorders) | 0 (0) | 2 (5)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less